CLINICAL TRIAL: NCT05358704
Title: Preoperative ChemoRadiation And FOLFOXIRI To Escalate Complete Response for Rectal Cancer (CRAFTER)
Brief Title: Preoperative ChemoRadiation And FOLFOXIRI for Rectal Cancer (CRAFTER) for Rectal Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: no slots available
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Salma Jabbour, MD, Professor of Radiation Oncology and Vice Chair, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072202; Pro2022000098 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Cancer of Rectum
Keywords: Cancer of Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; Capecitabine; Radiation; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Intervention Model Description: A single arm, open label, multi-institutional, Phase II trial of chemoradiation (CRT) followed by FOLFOXIRI for T3/T4 or lymph node positive rectal adenocarcinoma using a total neoadjuvant therapy (TNT) approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of drugs prior to surgery (Experimental): Receive the experimental combination of drugs (chemoradiation (capecitabine and radiation) + FOLFOXIRI (Oxaliplatin, leucovorin, irinotecan, and fluorouracil) prior to surgery and undergo laboratory tests and study procedures on specified days during the study period, complete end of study evaluations and tests, and participate in post-study follow up every three months for three to four years. The time in the study will take approximately four - six hours during pre-study, study and end of study visits.
  Interventions: Drug: combination of drugs (chemoradiation (capecitabine and radiation) + FOLFOXIRI (Oxaliplatin, leucovorin, irinotecan, and fluorouracil)

INTERVENTIONS:
Drug: combination of drugs (chemoradiation (capecitabine and radiation) + FOLFOXIRI (Oxaliplatin, leucovorin, irinotecan, and fluorouracil) — To evaluate the safety and preliminary efficacy of Preoperative ChemoRadiation and FOLFOXIRI To Escalate Complete Response for Rectal Cancer patients. receive the experimental combination of drugs (chemoradiation (capecitabine and radiation) + FOLFOXIRI (Oxaliplatin, leucovorin, irinotecan, and fluorouracil) and undergo laboratory tests and study procedures on specified days during the study period, complete end of study evaluations and tests, and participate in post-study follow up every three months for three to four years.
  Other Names: prior to surgery

SUMMARY:
To evaluate the safety and preliminary efficacy of Preoperative ChemoRadiation and FOLFOXIRI and to Escalate Complete Response for Rectal Cancer patients.Go through laboratory and medical tests to verify eligibility to enter the study, receive the experimental combination of drugs (chemoradiation (capecitabine and radiation) + FOLFOXIRI (Oxaliplatin, leucovorin, irinotecan, and fluorouracil) prior to surgery and undergo laboratory tests and study procedures on specified days during the study period, complete end of study evaluations and tests, and participate in post-study follow up every three months for three to four years. The time in the study will take approximately four to six hours during pre-study, study and end of study visits.

DETAILED DESCRIPTION:
Treatment will continue until participants experiences disease progression, unacceptable toxicity or withdraws consent and will include chemoradiation (28 days) followed by FOLFOXIRI x 8 cycles (16 weeks). A cycle is defined as an interval of fourteen days, except for Cycle 1 spanning fourteen days which includes eight cycles of FOLFOXIRI treatment prior to surgery. For participants experiencing unacceptable FOLFOXIRI or chemoradiation related toxicity, yet obtaining therapeutic benefit, participants will be allowed to continue treatment, if well tolerated at the discretion of the investigator.

Upon discontinuation of study treatment, participants will receive safety follow-up assessments approximately 30 and 90 days later. Once the 90-day safety follow-up is complete, participants will enter the survival follow-up period where they will continue to be followed approximately every three months until death, withdrawal of consent, or overall study completion. Patients will be followed for survival for 36 months from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Age 18 years or greater
* Be fully active, able to carry on all pre-disease performance without restriction or Restricted in physically strenuous activity but able to carry out work of a light or sedentary nature (e.g., light house work, office work)
* Pathologically proven diagnosis of adenocarcinoma of the rectum (located up to 15 cm from the anal verge). Diagnosis of rectal adenocarcinoma must be obtained by biopsy technique that does not completely excise the lesion (e.g., fine needle aspiration, core needle biopsy)
* Clinically determined to be stage T3 or T4, N0-N2, and M0
* Contrast-enhanced imaging of the abdomen by CT; MRI rectal protocol; Chest x-ray (or CT) of the chest All within 56 days prior to registration to exclude distant metastases and provide local tumor stage
* Adequate bone marrow function
* Adequate renal and liver function
* No active second cancers
* Be willing and able to comply with all aspects of the protocol
* Female patients of childbearing potential should have a negative pregnancy test within 72 hours prior to receiving the first dose of study medication
* Female patients of childbearing potential should be willing to use two methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Male patients should agree to abstinence or use of an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Zubrod Performance Status 0-2
* CBC/differential obtained within 28 days prior to registration on study, with adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,200 cells/mm3 Platelets ≥ 100,000 cells/mm3 Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable)
* Adequate hepatic function within within 28 days before registration on this study:

total bilirubin must be ≤ ULN (upper limit of normal) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and AST and ALT must be ≤3 x ULN for the lab If AST and/or ALT is ≥ ULN but ≤ 3 x ULN, serologic testing for Hepatitis B and C must be performed and results for viral infection must be negative

* Adequate renal function within 28 days before randomization defined as serum creatinine ≤ 1.5 x ULN for the lab or calculated creatinine clearance > 30 mL/min
* International normalized ratio of prothrombin time (INR) within 28 days before randomization must be ≤ ULN for the lab. Patients who are therapeutically treated with an agent such as warfarin may participate if they are on a stable dose and no underlying abnormality in coagulation parameters exists per medical history
* Acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease must:

Have a CD4 count ≥ 200 cells/μL within 30 days before randomization Be on a stable regimen of antiretroviral therapy Have no evidence of opportunistic infection

Exclusion Criteria:

* Age less than 18 years
* Pregnant or breastfeeding women
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of three years
* Prior systemic chemotherapy for colorectal cancer; note that prior chemotherapy for a different cancer is allowed.
* Prior radiotherapy to the region of your present study cancer that would result in overlap of radiation therapy fields
* Severe, active comorbidity, defined as follows:

Unstable angina and/or congestive heart failure requiring hospitalization within the last twelve months Transmural myocardial infarction within the last six months Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects Acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive Evidence of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake Known, existing uncontrolled coagulopathy. Patients on therapeutic anticoagulation may be enrolled provided that they have been clinically stable on anti-coagulation for at least two weeks

* Evidence of grade two or greater peripheral neuropathy
* Major surgery within 28 days of study enrollment
* Prior allergic reaction to oxaliplatin or capecitabine
* Any evidence of distant metastases
* A synchronous primary colon carcinoma
* Lack of physical integrity of the gastrointestinal tract (i.e., severe Crohn's disease that results in malabsorption; significant bowel resection that would make one concerned about the absorption of capecitabine) or malabsorption syndrome that would preclude feasibility of oral chemotherapy (capecitabine)
* Participation in any investigational drug study within 28 days of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Positron emission tomography (PET) | Four Years
  Standard tumor measurements using various scan studies. Scans are to be completed at each restaging time point. Participants will have cancer scan assessments every twelve weeks. Positron emission tomography (PET); Computed tomography (CT)can be used on this trial for response evaluation criteria in solid tumors (RECIST) measurements and can be used interchangeably with conventional Computed tomography (CT).

SECONDARY OUTCOMES:
Magnetic resonance imaging (MRI) | Four Years
  Standard tumor measurements using various scan studies. Scans are to be completed at each restaging time point.

OTHER OUTCOMES:
Computed tomography (CT) Scan of Chest, Abdomen and Pelvis (CT C/A/P) | Four Years
  Measurable lesions are defined as those that can be accurately measured in at least one dimension. This guideline has defined measurability of lesions on Computed tomography (CT) scan based on the assumption that Computed tomography (CT) slice thickness is 5 mm or less. If Computed tomography (CT) scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness each restaging time point.
Computed tomography (CT) | Four Years
  Measurable lesions are defined as those that can be accurately measured in at least one dimension. Malignant lymph nodes to be considered pathologically enlarged and measurable, a lymph node must be >15 mm in short axis when assessed by Computed tomography (CT) scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.
Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Four Years
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used for tumor measurements. Imaging for response assessment will be obtained before the initiation of conditioning (no more than four weeks prior to apheresis) and at the six-week follow up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Jabbour, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey; Patrick M Boland, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - RWJBarnabas Health - Monmouth Medical Center, Lakewood, New Jersey
  - RWJBarnabas Health - Saint Barnabas Medical Center, Livingston, Livingston, New Jersey
  - Rutgers, The State University of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, Somerset, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No